CLINICAL TRIAL: NCT00066092
Title: Randomized, Double-Blind Study of Peripheral Blood Progenitor Cell (PBPC) Mobilization by Pegfilgrastim or Filgrastim for Autologous Transplantation in Subjects With Hodgkin's or Non-Hodgkin's Lymphoma.
Brief Title: Pegfilgrastim PBPC Mobilization Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20020112; NCT00060229 (obsolete NCT alias)
Record Dates: First submitted 2003-08-04; First posted 2003-08-05 (Estimated); Last update posted 2008-02-28 (Estimated); Status verified 2008-02

CONDITIONS: Lymphoma; Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Hematology; Oncology
Keywords: PBPC transplant; Hodgkin's Disease; Non-Hodgkin's Lymphoma; NHL; mobilization
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Neoplasms | interventions — pegfilgrastim; Filgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Pegfilgrastim 6 mg (Experimental): Pegfilgrastim 6 mg given once for PBPC mobilization
  Interventions: Drug: pegfilgrastim 6 mg
- Pegfilgrastim 12 mg (Experimental): Pegfilgrastim 12 mg given once for PBPC mobilization
  Interventions: Drug: pegfilgrastim 12 mg
- filgrastim (Active Comparator): Filgrastim given daily for PBPC mobilization
  Interventions: Drug: filgrastim

INTERVENTIONS:
Drug: pegfilgrastim 12 mg — Pegfilgrastim 12 mg given once for PBPC mobilization
  Arms: Pegfilgrastim 12 mg
Drug: filgrastim — Filgrastim given daily for PBPC mobilization
  Arms: filgrastim
Drug: pegfilgrastim 6 mg — Pegfilgrastim 6 mg given once for PBPC mobilization
  Arms: Pegfilgrastim 6 mg

SUMMARY:
This is a randomized, double-blind, multi-center study to assess the safety and effectiveness of using a single subcutaneous (under the skin) injection of pegfilgrastim or daily subcutaneous injections of Filgrastim to mobilize stem cells for autologous transplantation in patients with Hodgkin's or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
This is a research study for Hodgkin's Disease and Non-Hodgkin's Lymphoma (NHL) patients who will receive high-dose chemotherapy with autologous peripheral blood stem cell (PBSC or PBPC) transplant. The chemotherapy doses are high enough to severely suppress the bone marrow (where blood cells are made) and cause very low blood counts. A collection of stem cells (very young blood cells) followed by reinfusion to restore blood counts will be done to stimulate recovery of your blood counts. This procedure is called leukapheresis. Giving growth factors to patients is a method to increase the number of PBPC that can be collected during leukapheresis. This process of giving growth factors to patients is called mobilization (moving cells from the bone marrow to the peripheral blood where they can be collected). The purpose of this study is to determine if pegfilgrastim, an investigational drug, can safely and effectively mobilize stem cells. Filgrastim (also known as NEUPOGEN® or G-CSF) is approved by the FDA for stem cell mobilization. Pegfilgrastim is a modified version of Filgrastim that is longer acting.

ELIGIBILITY:
* Hodgkin's or non-Hodgkin's lymphoma patients suitable for an autologous PBPC transplant - No previous bone marrow or PBPC transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2003-04; Primary Completion 2004-03 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
CD34+ collection during the collection phase | 10 days

SECONDARY OUTCOMES:
Time to ANC and platelet engraftment post-transplant | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20020112.pdf